CLINICAL TRIAL: NCT00236990
Title: A Double-Blind, Randomized, Placebo-Controlled Trial of ELMIRON (Pentosan Polysulfate Sodium) for the Treatment of Chronic Non-Bacterial Prostatitis
Brief Title: An Effectiveness and Safety Study of ELMIRON (Pentosan Polysulfate Sodium) for the Treatment of Chronic Non-Bacterial Inflammation of the Prostate Gland
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Collaborators: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004687
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Prostatitis
Keywords: prostatitis; Elmiron; pentosan polysulfate sodium
MeSH Terms: conditions — Prostatitis | interventions — Pentosan Sulfuric Polyester

ARMS (1):
- 001 (Experimental): pentosan polysulfate sodium
  Interventions: Drug: pentosan polysulfate sodium

INTERVENTIONS:
Drug: pentosan polysulfate sodium

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of ELMIRONÂ® in the treatment of chronic non-bacterial inflammation of the prostate gland.

DETAILED DESCRIPTION:
The objective of this randomized, double-blind, placebo-controlled study is to determine the effectiveness and safety of ELMIRON® 100 mg three times per day for 12 weeks, as compared with placebo, in patients with chronic non-bacterial inflammation of the prostate gland. Safety evaluations will be assessed throughout the study. The hypothesis of the study is that ELMIRON® will be more effective than placebo, as based on the change in the total National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) score from baseline to the final visit (Week 12) and is generally well-tolerated. Patients will receive oral ELMIRON® 100 mg three times per day orally or matching placebo three times per day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic non-bacterial prostatitis/chronic pelvic pain syndrome
* symptoms of discomfort or pain in the perineal and/or pelvic region (lower abdomen) for at least three of the last six months for which there is no recognized cause
* symptoms persist despite treatment with antibiotics for non-bacterial prostatitis in the past six months.

Exclusion Criteria:

* Clinically significant medical problems or other organ abnormalities
* psychiatric disorders
* urinary tract infection during the last three months
* history of bladder, urethral or prostate cancer
* Prostate Specific Antigen (PSA) greater than or equal to 4 ng/mL
* diagnosis or treatment for genital herpes or herpes flare within the last year.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The change in total NIH-CPSI score from baseline to Week 12

SECONDARY OUTCOMES:
Participant-reported Global Response Assessment at Week 12. Brief Male Sexual Function Index at Weeks 4, 8, and 12. Pelvic Pain Urgency and Frequency symptom scale at Weeks 4, 8, and 12.

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- See also: An Effectiveness and Safety Study of ELMIRON� (Pentosan Polysulfate Sodium) for the Treatment of Chronic Non-Bacterial Inflammation of the Prostate Gland — http://download.veritasmedicine.com/PDF/CR004687_CSR.pdf